CLINICAL TRIAL: NCT01158794
Title: Genes Influencing Iron Overload State
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GENIOS
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Sickle Cell Disease; Thalassemia; Marrow Aplasia
Keywords: Iron overload; Blood Transfusion
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The total volume of blood transfused (in ml/kg) will be collected and stored in the study database. Cumulative transfused blood volume (in ml/kg) will be captured. Serum samples will be stored frozen at -20°C until the time of analysis. In addition to the protocol-specific testing of specimens, study participants will be offered the option of allowing any leftover purified DNA, serum, or blood cells to be saved or shared for future analyses. Leftover purified genomic DNA, serum, and blood cells from subjects enrolled in the GENIOS protocol will be de-identified prior to storage or any future testing and/or sharing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: Participants with sickle cell disease and transfusional iron-overload, and non-sickle cell disease (thalassemia major, cancer patients, etc.) and iron overload. Participants with iron overload, defined as too much iron in the body as a consequence of too many blood transfusions.

SUMMARY:
Iron overload, which can be defined operationally as too much iron in the body, develops as a consequence of too many blood transfusions given, or due to genetic defects hereditary hemochromatosis). Iron accumulates in several organs in the body, such as the heart, liver, endocrine glands (pancreas, thyroid, etc.), and spleen. Excessive iron can damage organs and may even cause death. Iron overload needs to be appropriately monitored and treated to avoid unnecessary morbidity and mortality.

The present study, GENIOS, proposes to test prospectively the hypothesis that genetic modifiers influence the iron overload status of patients receiving transfusions. To test this hypothesis, the study will perform genetic studies to investigate possible genetic influences for iron accumulation in the body and will study iron accumulation not only in the liver, but also in the heart, pancreas, kidneys, and spleen. In addition: the study will investigate if these same genes have any role during treatment of iron overload, in other words, if certain genetic mutations will influence how iron exits the body. This study will also investigate how substances that are known to control the trafficking of iron in and out of the body and its damaging effects to the tissues (hepcidin and non transferrin-bound iron) are linked to the accumulation of iron in the heart and liver. Iron in the body will be measured by R2*MRI and no liver biopsies will be required. Genetic studies will be done by specialized tests using peripheral blood DNA.

Iron accumulates differently in different people and in different organs of the body. Some people accumulate iron faster than others, even when receiving the same number of blood transfusions

DETAILED DESCRIPTION:
This study will focus on the following primary objective:

* To investigate the association of GSTM1 gene deletion and liver iron concentration in patients with sickle cell disease and transfusional iron-overload.

The Secondary Objectives of the study are:

* To explore the role of other iron metabolism-associated candidate genes on liver iron concentration of sickle cell patients with transfusional iron-overload.
* To explore the role of GSTM1 genotypes and other iron metabolism-associated candidate genes on maintenance and decline of liver iron concentration of patients with sickle cell disease and transfusional iron-overload.
* To explore the role of GSTM1 genotypes and other iron metabolism-associated candidate genes on increase, maintenance, and decline of iron concentration in the heart, pancreas, kidneys, and spleen of patients with sickle cell disease and transfusional iron overload.
* To explore the role of GSTM1 gene deletion and other iron metabolism-associated candidate genes on increase, maintenance, and decline of iron concentration in the liver, heart, pancreas, kidneys, and spleen of non-sickle cell patients with transfusional iron-overload.
* To explore the relationship between Non-Transferrin Bound Iron (NTBI), hepcidin, organ function, and iron increase, maintenance, and decline in the liver, heart, pancreas, kidneys, and spleen of patients with transfusional iron overload.

ELIGIBILITY:
Inclusion Criteria:

* History of ≥ 12 lifetime erythrocyte transfusions who have not yet initiated treatment to unload iron (iron chelation or therapeutic phlebotomy), or
* History of ≥ 12 lifetime erythrocyte transfusions who have initiated treatment to unload iron, but had liver iron content measurement (by R2*MRI) within 3 months prior to initiation of iron unloading treatment

Exclusion Criteria

* Known contraindication to performance of MRI (e.g.: presence of MRI-incompatible ferromagnetic material in the body)
* Prior participation on the St. Jude MRIRON protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be patients who receive medical care at St. Jude Children's Research Hospital and have developed iron overload secondary to multiple transfusions. Patients will be approached during regular outpatient visits and will be invited to participate in this study if they meet the inclusion/exclusion criteria and consent to participate in the study. Non-sickle cell patients with transfusional iron overload includes patients with thalassemia, bone marrow failure syndromes, and patients who have received multiple blood transfusions due to marrow aplasia secondary to the use of chemotherapeutic agents. About 40 participants with sickle cell disease are targeted. About 10 participants with non-sickle cell disease are targeted.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09-21 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
This study will measure genetic modifiers influencing the iron overload status of patients receiving transfusions. | Once, at participant enrollment
  This study will measure the association between GSTM1 gene deletion and other candidate genes and the accumulation and clearance of body iron.

SECONDARY OUTCOMES:
To explore the role of other iron metabolism-associated candidate genes on liver iron concentration of sickle cell patients with transfusional iron-overload. | Once, at participant enrollment
To explore the role of GSTM1 genotypes and other iron metabolism-associated candidate genes on maintenance and decline of liver iron concentration of patients with sickle cell disease and transfusional iron-overload. | Once at baseline compared to 3 years after participant enrollment
Explore the role of GSTM1 genotypes and other iron metabolism-associated candidate genes on increase, maintenance, and decline of iron concentration patients with sickle cell disease and transfusional iron overload. | Once at baseline compared to 3 years after participant enrollment
  Decline of iron concentration is in the heart, pancreas, kidneys, and spleen.
Explore the role of GSTM1 gene deletion and other iron metabolism-associated candidate genes on increase, maintenance, and decline of iron concentration of non-sickle cell patients* with transfusional iron-overload. | Once at baseline compared to 3 years after participant enrollment
  Decline of iron concentration in the liver, heart, pancreas, kidneys, and spleen of non-sickle cell patients with transfusional iron-overload.
Explore the relationship between Non-Transferrin Bound Iron (NTBI), hepcidin, organ function, and iron increase, maintenance, and decline in the liver, heart, pancreas, kidneys, and spleen of patients with transfusional iron overload. | Once at baseline compared to 3 years after participant enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols